CLINICAL TRIAL: NCT03348605
Title: Descriptive Study of Receptive Fields in Lower Limb Amputees and the Effect of a Related Stimulation System on Selected Gait Parameters
Brief Title: Descriptive Study of Receptive Fields in Lower Limb Amputees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rehaklinik Bellikon (Other)
Collaborators: Cort X Sensorics GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 01_2017; 2017-01621 (Other: SNCTP (Swiss National Clinical Trials Portal))
Record Dates: First submitted 2017-10-30; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Lower Limb Amputation Below Knee (Injury)
Keywords: Amputation; Phantom Pain; Gait analysis
MeSH Terms: conditions — Wounds and Injuries; Phantom Limb

STUDY DESIGN:
Intervention Model Description: The primary outcomes are the changes in size and position over time and their timed occurrence after the amputation of these receptive fields as well as the inter-/intratester reliability in their detection.
  The secondary outcomes are the change in selected gait parameters and phantom sensations through the application of the stimulating system ("Phantom Stimulator" (Cort X Sensorics, Spaichingen, Germany)).
  The primary outcome is of mere descriptive nature. Therefore, no control group is created and the participants are not blinded or randomized.
  For the secondary outcomes, every tested subject serves as its own control (cross over). The gait analysis as well as the questionnaire are performed three times. The two measurements after the first familiarization measurements are performed in a randomized order.
Who Masked: Participant
Masking Description: As this study is described as single blinded, the only entity of the trial not aware of the group or sequence of the participant is the participant itself.
  The other personell involved in the trial needs to be aware of the position of the participant within the study so to apply the right measures.
  In this case the participant is unaware of the fact whether his stimulation system is turned on or off.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First setting ON (Other): This arm performs the Gait analysis the first time after the familiarization phase with the stimulator in the modality ON. The second time the gait analysis is performed in the OFF modality.
  Interventions: Device: Phantom Stimulator, Cort X Sensorics, Spaichingen, Germany
- First setting OFF (Other): This arm performs the Gait analysis the first time after the familiarization phase with the stimulator in the modality OFF. The second time the gait analysis is performed in the ON modality.
  Interventions: Device: Phantom Stimulator, Cort X Sensorics, Spaichingen, Germany

INTERVENTIONS:
Device: Phantom Stimulator, Cort X Sensorics, Spaichingen, Germany — This system consists of a pressure sensing insole connected to regular TENS-Electrode patches which are applied to the receptive fields of the patients (evoking the sensation of heel and forefoot). The individually adjusted stimulation intensity on the systems regulatory box through a socked screw is set at the beginning of the testing phase, and not changed anymore.
  The current is applied to mimic the roll-off-sensation while walking. This is done by locating two sets of electrodes on the receptive fields representing the heel and the ball of the foot respectively. Now the current is applied in an alternating manner coordinated with the walking of the participant. The coordination is made able through the pressure sensing insole.

SUMMARY:
It has been observed that patients subjected to amputations develop so called receptive fields, which time of occurrence and localization over time are yet not examined systematically.

This clinical trial aims to investigate the reliability in detecting these receptive fields as well as their incidence and changes over time.

Further it aims to evaluate the acute effect of a stimulating system ("Phantom Stimulator" (Cort X Sensorics, Spaichingen, Germany)) on selected gait parameters measured tough a gait analysis system ("OprtoGait" (Microgate, Bolzano, Italy)) as well as on phantom sensations measured through a questionnaire.

DETAILED DESCRIPTION:
It has been observed that patients subjected to amputations develop so called receptive fields, which time of occurrence and localization over time are yet not examined systematically.

A receptive field is defined as skin area anywhere on the same side of the body as the amputation, which when stimulated by others, causes phantom sensations in the amputated extremity.

This clinical trial aims to investigate the reliability in detecting these receptive fields as well as their incidence and changes over time.

Further it aims to evaluate the acute effect of the stimulating system ("Phantom Stimulator" (Cort X Sensorics, Spaichingen, Germany)) on selected gait parameters measured tough a gait analysis system ("OprtoGait" (Microgate, Bolzano, Italy)) as well as on phantom sensations measured through a questionnaire.

ELIGIBILITY:
1. Inclusion criteria for descriptive study:

   a. Lower limb amputation (independently of side or height of amputation)
2. Inclusion criteria for Phantom stimulator:

   1. Receptive fields present at testing day 31 (last regular assessment of the receptive fields)
   2. Lower limb amputation below the knee (if both sides the system is applied to the dominant side).
3. Exclusion criteria:

   1. Implanted devices (defibrillator or pacemaker)
   2. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Description of receptive Fields Size in cm2 | 4-5 Weeks (7 hours)
  The primary outcomes are the changes in size over time. Here the size is described in cm2. The Fields size will be recorded by drawing them on the skin with eyeliner and subsequently taking photos.
  Later, these photos are analysed with the computer program Photoshop.
Description of receptive Fields Position in % overlapping from first measurement | 4-5 Weeks (7 hours)
  The primary outcomes are the changes in Position over time. Here the position is described in % overlapping with respect to the first measurement.
  The Fields position will be recorded by drawing them on the skin with eyeliner and subsequently taking photos. Later, these photos are put together and compared with the computer program Photoshop.

SECONDARY OUTCOMES:
Change in gait parameters through Phantom Stimulator | 1/2 Day (3 hours)
  The secondary outcomes are the change in selected gait parameters through the application of the stimulating system ("Phantom Stimulator" (Cort X Sensorics, Spaichingen, Germany)).
  These parameters are measured with the gait analysis system Optogait. The selected parameters are step length (cm), width (cm), cadence (steps/min) and speed (m/s).
Change in phantom sensations through Phantom Stimulator | 1/2 Day (3 hours)
  The secondary outcomes are the change in phantom sensations through the application of the stimulating system ("Phantom Stimulator" (Cort X Sensorics, Spaichingen, Germany)).
  These changes are measured through a questionnaire witch uses the Visual Analogue Scale (values from 1 - 10).

CONTACTS AND LOCATIONS:
Overall Officials: Marion Grögli, Dr. med., Principal Investigator — Reahklinik Bellikon
Locations (1):
- Rehaklinik Bellikon, Bellikon, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No
IPD is used only internally the study concerning the Phantom Stimulator (Cort X Sensorics, Spaichingen Germany). The IPD is shared with the responsible investigative parties of the Rehaklinik Bellikon only.
  It will be available to the participant after completion of the study. The data obtained from the Study results in a publication after completion of the study.

REFERENCES:
- See also: Website of study site — http://www.rehabellikon.ch/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT03348605/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT03348605/ICF_001.pdf